CLINICAL TRIAL: NCT04102956
Title: Human Urinary Kallidinogenase Improve Short Term Motor Functional Outcome by Reducing the Corticospinal Tract Damage in Acute Ischemia Stroke Patients
Brief Title: Human Urinary Kallidinogenase Improve Short Term Motor Functional Outcome of Acute Ischemia Stroke Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Second Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, liuxiaoyun, Deputy Director of Neurology Department, The Second Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-P023
Record Dates: First submitted 2019-09-18; First posted 2019-09-25 (Actual); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke | interventions — Kallikreins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kallikrein+Standard treatment group (Experimental): The Kallikrein+Standard treatment group was given kallikrein through intravenous injection to treatment for 0.15 PNA/day+standard treatment medicine based on the guidelines for the treatment of acute ischemic stroke for 14 ± 5 days.
  Interventions: Drug: Kallikrein
- Standard treatment group (No Intervention): The Standard treatment group was only given standard treatment medicine based on the guidelines for the treatment of acute ischemic stroke for 14 ± 5 days.

INTERVENTIONS:
Drug: Kallikrein — HUK has been approved by China's State Food and Drug Administration as a state category I new drug for the treatment of stroke patients. Based on the available evidence, HUK injection ameliorates neurological deficits and improves long-term outcomes.
  Other Names: Human urinary kallidinogenase
  Arms: Kallikrein+Standard treatment group

SUMMARY:
Acute cerebral infarction is a common type of ischemic stroke, causing brain dysfunction in patients with high morbidity and disability. With the changes in people's diet, lifestyle patterns and population aging, the incidence of acute cerebral infarction has increased year by year, which has become an important cause of disability and death in middle-aged and elderly patients. The human urinary kallidinogenase (HUK) was used in China in the management of acute ischemic stroke (AIS) in recent years. However, the mechanism of HUK on AIS has not been systematically investigated. This study aimed to assess the effect of HUK on motor functional outcome and relative corticospinal tract recovery in the patients with AIS. Diffusion tensor imaging(DTI) and diffusion tensor tractography(DTT) have all been used to observe features of cerebral white matter fibrous structures. In addition, diffusion tensor tractography which is used to trace fiber bundle and evaluate white matter fiber bundle integrity and direction is the only non-invasive imaging method to display the corticospinal tract in vivo.

DETAILED DESCRIPTION:
A total of 80 AIS patients with the unilateral corticospinal tract damage who were matched for inclusion criterion were enrolled in this randomized controlled trial. The HUK group was administered with HUK and standard treatment(general treatment for anti-platelet, lipid-lowering and improving circulation,etc.), the control group received only standard treatment. Kallikrein+Standard Treatment Group (general Treatment for anti-platelet, lipid-lowering and improving circulation,etc.) and Standard Treatment Group were randomly selected.

At admission and discharge, National Institute of Health Stroke Scale(NIHSS), Barthel Index(BI), muscle strength were scored; The DTI were performed and DTT were utilized to reconstruct corticospinal tract to observe its direction and appearance changes then to evaluate the integrity and impairment degree of the corticospinal tract which was divided into four grades according to DTT presented compression, deformation, or rupture. Fractional anisotropy(FA) and apparent diffusion coefficient(ADC) of infarct region and corresponding contralateral normal regions were measured.

Blood samples were collected to test serum myelin basic protein(MBP) and vascular endothelial growth factor (VEGF) by enzyme-linked immunosorbent assay (ELISA). The primary endpoint is the short-term motor function prognosis of the AIS patients, we also evaluated the recovery of corticospinal tract and the serum MBP and VEGF changes during treatment in two groups.

ELIGIBILITY:
Inclusion Criteria:

18 years old ≤ age <80 years old; Within 72 hours of onset; Diagnosed as acute cerebral infarction, and confirmed by magnetic resonance imaging as an acute infarct in the unilateral corticospinal tract; The patient's onset muscle strength grade <4; No history of cerebral infarction or residual physical activity disorder; No other intracranial lesions; Patients or their legal representatives voluntarily Sign the informed consent form;

Exclusion Criteria:

Intracranial hemorrhagic disease: cerebral hemorrhage, subarachnoid hemorrhage, etc.; Transient ischemic attack; Intravenous thrombolysis and interventional thrombectomy; Serious physical illness affects limb movement before enrollment ; Apply other drugs with nutritional nerves and regeneration during the study period; Unstable vital signs, severe liver and kidney diseases or malignant tumors; Incomprehensible or incapable of obeying the research procedure or being unable to follow up due to mental illness, cognitive or emotional disorders;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyun Liu, Prf., Principal Investigator — The Second Hospital of Hebei Medical University
Locations (1):
- Second hospital of hebei medical university, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Li P, Lu H, Shi X, Yan J, Zhou L, Yang J, Wang B, Zhao Y, Liu L, Zhu Y, Xu L, Yang X, Su X, Yang Y, Zhang T, Guo L, Liu X. Protective effects of human urinary kallidinogenase against corticospinal tract damage in acute ischemic stroke patients. Neuroreport. 2024 May 8;35(7):431-438. doi: 10.1097/WNR.0000000000002028. Epub 2024 Mar 12. PMID 38526971

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kallikrein+Standard Treatment Group | Standard Treatment Group
Started | 42 | 38
Completed | 42 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kallikrein+Standard Treatment Group | Standard Treatment Group | Total
Number analyzed (Participants) | 42 | 38 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.762 (11.096) | 60.789 (9.376) | 58.675 (10.4479)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 30 | 22 | 52
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hypertension (number, %) [Count of Participants; unit: Participants]
  Have hypertension | 33 | 29 | 62
  Without hypertension | 9 | 9 | 18
Diabetes (number, %) [Count of Participants; unit: Participants]
  Diabetes | 15 | 13 | 28
  Without diabetes | 27 | 25 | 52
Coronary heart disease (number, %) [Count of Participants; unit: Participants]
  With coronary heart disease | 3 | 5 | 8
  Without coronary heart disease | 39 | 33 | 72
Hyperhomocysteinemia (number, %) [Count of Participants; unit: Participants]
  Hyperhomocysteinemia | 18 | 14 | 32
  without hyperhomocysteinemia | 24 | 24 | 48
Previous history of cerebral infarction (number, %) [Count of Participants; unit: Participants]
  Previous history of cerebral infarction | 7 | 7 | 14
  Without the history of cerebral infarction | 35 | 31 | 66
Smoking and drink (number, %) [Count of Participants; unit: Participants]
  Smoking and drink | 25 | 16 | 41
  No history of smoking or drinking | 17 | 22 | 39
Muscle strength at admission，Median (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — The 6-level muscle strength recording method of 0-5 levels is used. Level 0 means no muscle contraction, and level 5 means normal muscle strength.
  units on a scale | 2 [1 to 3] | 2 [1 to 3] | 2 [1 to 3]
NIHSS score at admission ( Mean±SD) [Mean (Standard Deviation); unit: units on a scale] — The National Institute of Health Stroke Scale(NIHSS) ranges from 0 to 42, with the higher the score, the more severe the nerve damage.
  units on a scale | 9.21 (3.258) | 8.05 (3.196) | 8.66 (3.261)
BI index at admission，Median (IQR) [Median (Inter-Quartile Range); unit: units on a scale] — Barthel Index(BI) ranges from 0 to 100 points, the higher the score, the stronger the self-care ability.
  units on a scale | 25 [20 to 40] | 25 [20 to 40] | 25 [20 to 40]
FA value at admission ( Mean±SD) [Mean (Standard Deviation); unit: units on a scale] — The Fractional Anisotropy (FA) value is used to express the anisotropy, which indicates the anisotropic component of water molecules accounts for the total value of diffusion tensor,and ranges from 0 to 1, the closer the value is to 1, the better the fiber bundle integrity. Population: 78 taken the DTI imaging at admission (40 in the Kallikrein+Standard treatment group and 38 in the Standard treatment group)
  units on a scale
    number analyzed (Participants) | 40 | 38 | 78
    (all) | 0.441 (0.055) | 0.427 (0.044) | 0.436 (0.484)
ADC value at admission ( Mean±SD) [Mean (Standard Deviation); unit: m㎡/s] — The ADC value of normal brain tissue is in the range of 0.7-0.9×10﹣³m㎡/s. When the brain tissue is acutely affected, it is mostly decreased, and it is mostly increased in subacute or chronic disease. The upper and lower limits of abnormal changes in ADC value are 0.4-2.5×10﹣³m㎡/s. Population: Measure Analysis Population Description: 78 taken the DTI imaging at admission (40 in the Kallikrein+Standard treatment group and 38 in the Standard treatment group).
  m㎡/s
    number analyzed (Participants) | 40 | 38 | 78
    (all) | 0.811 (0.209) | 0.847 (0.081) | 0.831 (0.162)
The grade of the severity of corticospinal tract injury ( number, %) [Count of Participants; unit: Participants] — The severity of the corticospinal tract injury evaluated according to DTT presented compression, deformation, or rupture was classified as: Grade 1 refers to complete corticospinal tract; Grade 2 refers to slight corticospinal injury less than 50%. Grade 3 refers to moderate corticospinal tract injury between 50%~75%; Grade 4 refers to severe corticospinal tract injury, almost interrupted more than 75%.
  Participants
    Grade 1 | 6 | 6 | 12
    Grade 2 | 20 | 9 | 29
    Grade 3 | 13 | 16 | 29
    Grade 4 | 3 | 7 | 10
Intracranial arterial stenosis ( number, %) [Count of Participants; unit: Participants]
  Intracranial arterial stenosis | 20 | 14 | 34
  Without intracranial arterial stenosis | 22 | 24 | 46
VEGF Median (IQR) (pg/ml) [Median (Inter-Quartile Range); unit: pg/ml] — Population: Among the enrolled 80 subjects, 59 taken the blood samples (33 in the Kallikrein+Standard treatment group and 26 in the Standard treatment group) to teste the concentrations of VEGF and MBP.
  pg/ml
    number analyzed (Participants) | 33 | 26 | 59
    (all) | 22.43 [10.02 to 50.43] | 22.56 [16.06 to 55.24] | 22.46 [10.54 to 51.97]
MBP Median (IQR) (pg/ml) [Median (Inter-Quartile Range); unit: pg/ml] — Population: Among the enrolled 80 subjects, 59 taken the blood samples (33 in the Kallikrein+Standard treatment group and 26 in the Standard treatment group) to teste the concentrations of VEGF and MBP.
  pg/ml
    number analyzed (Participants) | 33 | 26 | 59
    (all) | 0.42 [0.23 to 0.80] | 0.64 [0.15 to 1.36] | 0.56 [0.23 to 1.08]

OUTCOME MEASURES:

1. Primary Outcome: Myelin Basic Protein (MBP) Comparison Between the Two Groups Before and After Treatment
Description: The effect of Kallikrein on myelin basic protein (MBP) was determined by comparing the changes of MBP before and after treatment between the Kallikrein+Standard treatment group and the standard treatment group.
Time Frame: before (baseline) and after treatment (14 ± 5 days)
Population: Among the enrolled 80 subjects, 59 taken the blood samples (33 in the Kallikrein+Standard treatment group and 26 in the Standard treatment group) to test serum myelin basic protein(MBP) and vascular endothelial growth factor (VEGF).
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Kallikrein+Standard Treatment Group | Standard Treatment Group
Number analyzed (Participants) | 33 | 26
pg/ml
  Prior treatment | 0.42 [0.23 to 0.80] | 0.64 [0.15 to 1.36]
  After treatment | 0.41 [0.18 to 0.82] | 0.71 [0.27 to 1.35]

2. Primary Outcome: Comparison of Vascular Endothelial Growth Factor (VEGF) Before and After Treatment Between the Kallikrein+Standard Treatment Group and Standard Treatment Group
Description: The effect of Kallikrein on vascular endothelial growth factor (VEGF) was judged by comparing the changes of VEGF before and after treatment in the Kallikrein+Standard treatment group and the standard treatment group.
Time Frame: before (baseline) and after treatment (14 ± 5 days)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Kallikrein+Standard Treatment Group | Standard Treatment Group
Number analyzed (Participants) | 33 | 26
ng/ml
  Prior treatment | 22.42 [10.25 to 50.43] | 22.56 [16.06 to 55.24]
  After treatment | 29.53 [17.31 to 59.68] | 22.91 [9.97 to 47.62]

3. Primary Outcome: Changes of Barthel Index(BI) Before and After Treatment in the Two Groups
Description: The Barthel Index(BI) is 0 to 100 points. The higher the score, the better the patient's motor function and behavior. The effect of Kallikrein on Barthel Index was judged by comparing the changes of Barthel Index before and after treatment in the Kallikrein+Standard treatment group and the standard treatment group.
Time Frame: before (baseline) and after treatment (14 ± 5 days)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Kallikrein+Standard Treatment Group | Standard Treatment Group
Number analyzed (Participants) | 42 | 38
score on a scale | 17.5 [10 to 30] | 12.5 [5 to 20]

4. Primary Outcome: Changes in Muscle Strength of the Kallikrein+Standard Treatment Group and the Standard Treatment Group Before and After Treatment
Description: Using the recording method of grade 6 muscle strength of 0-5 grade, grade 0 means no muscle contraction, grade 5 means normal muscle strength. The effect of Kallikrein on muscle strength was judged by comparing the changes of muscle strength before and after treatment in the Kallikrein+Standard treatment group and the standard treatment group.
Time Frame: before (baseline) and after treatment (14 ± 5 days)
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Kallikrein+Standard Treatment Group | Standard Treatment Group
Number analyzed (Participants) | 42 | 38
score on a scale | 1 [0 to 1] | 1 [1 to 2]

5. Primary Outcome: Changes of National Institute of Health Stroke Scale(NIHSS) Before and After Treatment in the Two Groups
Description: The NIHSS score is 0 to 42 points. The higher the score, the more severe the nerve damage. The change of NIHSS score is calculated as the value at the earlier time point minus the value at the later time point, that is, the value at the time of admission minus the value after the end of treatment, and then the comparison between groups is performed to obtain the current result.
Time Frame: before (baseline) and after treatment (14 ± 5 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kallikrein+Standard Treatment Group | Standard Treatment Group
Number analyzed (Participants) | 42 | 38
score on a scale | 2.88 (1.35) | 2.16 (1.59)

6. Primary Outcome: Change of Fractional Anisotropy Valuev Decline Rate† (FA Decline Rate†)
Description: The FA value is used to express the anisotropy, which indicates the anisotropic component of water molecules accounts for the total value of diffusion tensor,and ranges from 0 to 1, the closer the value is to 1, the better the fiber bundle integrity.
  †FA decline rate = (FA contralateral- FA ipsilateral) / FA contralateral， Used to compare the FA decline rate† of the two groups after treatment. A more substantial decrease of FA values is believed to represent the most severely ischemic tissue.
Time Frame: After 14 ± 5 days of treatment
Measure: Median (Inter-Quartile Range); unit: percentage of decline rate
Arm/Group | Kallikrein+Standard Treatment Group | Standard Treatment Group
Number analyzed (Participants) | 40 | 38
percentage of decline rate | 0.036 [-0.001 to 0.099] | 0.09 [0.05 to 0.16]

7. Primary Outcome: Change of Apparent Diffusion Coefficient Value Decline Rate‡（ADC Decline Rate‡）
Description: The ADC value of normal brain tissue is in the range of 0.7-0.9×10﹣³m㎡/s. When the brain tissue is acutely affected, it is mostly decreased, and it is mostly increased in subacute or chronic disease. The upper and lower limits of abnormal changes in ADC value are 0.4-2.5×10﹣³m㎡/s. ‡ ADC decline rate = (ADCcontralateral- ADCipsilateral) / ADCcontralateral；Used to compare the ADC decline rate‡ of the two groups after treatment. A more substantial decrease of ADC values is believed to represent the most severely ischemic tissue.
Time Frame: After 14 ± 5 days of treatment
Measure: Median (Inter-Quartile Range); unit: percentage of decline rate
Arm/Group | Kallikrein+Standard Treatment Group | Standard Treatment Group
Number analyzed (Participants) | 40 | 38
percentage of decline rate | -0.02 [-0.06 to 0.01] | 0.03 [-0.02 to 0.07]

ADVERSE EVENTS:
Time Frame: During the hospitalization of all participants within 14 ± 5 days
Description: No adverse events
Arm/Group | Kallikrein+Standard Treatment Group | Standard Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/38
Other Adverse Events (participants affected / at risk) | 0/42 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT04102956/ICF_001.pdf
  • Study Protocol (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT04102956/Prot_002.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT04102956/SAP_003.pdf